CLINICAL TRIAL: NCT06662123
Title: A Randomized, Phase I, Open-Label, Single-Dose Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of Subcutaneously and Intravenously Delivered Anifrolumab in Healthy Chinese Participants
Brief Title: Pharmacokinetic and Safety Study of Subcutaneous and Intravenous Anifrolumab Delivered in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D3465C00004
Record Dates: First submitted 2024-09-04; First posted 2024-10-28 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — anifrolumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Subcutaneous (Experimental)
  Interventions: Drug: Anifrolumab
- Intravenous (Experimental)
  Interventions: Drug: Anifrolumab

INTERVENTIONS:
Drug: Anifrolumab — Participants will receive a single SC or IV dose of anifrolumab at day 1
  Other Names: Saphnelo

SUMMARY:
This is a randomized, Phase I, open-label, single-dose study to evaluate the PK, safety, and tolerability of anifrolumab administered to male and female healthy Chinese participants aged 18 to 55 years. Approximately 24 participants, who fulfill the eligibility criteria, will be administered anifrolumab via SC route or IV route, and participants will be randomized to the two arms in a 1:1 ratio.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the PK, safety, and tolerability of a single dose of anifrolumab subcutaneously or intravenously administered to healthy Chinese participants aged 18 to 55 years. The primary study endpoints are PK standard endpoints. The secondary study endpoints are standard endpoints for safety assessment, including adverse events, serious adverse events, and clinical safety laboratory measurements. The participants must abstain from taking prescription or non-prescription drugs (including vitamins and dietary or herbal supplements) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) before the start of study intervention until completion of the follow-up visit, unless, in the opinion of the investigator and sponsor, the medication will not interfere with the study.

ELIGIBILITY:
Inclusion Criteria:

* Able to complete the follow-up visit as required by the protocol.
* Participant must be 18 to 55 years of age (both inclusive), at the time of signature of the ICF.
* A body mass index of ≥ 18.5 to ≤ 26.0 kg/m2 and body weight of at least 45 kg for females and 50 kg for males at screening.
* Capable of giving signed informed consent as described in Appendix A which includes compliance with the requirements and restrictions listed in the ICF and in this protocol.

Exclusion Criteria:

* History of malignancy with some exceptions
* History of alcohol or drug abuse within the past 2 years.
* Any significant disease, disorder, or finding that may significantly increase the risk to the participant because of participation in the study, affect the ability of the participant to participate in the study, or impair interpretation of the study data.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2024-10-21 (Actual); Primary Completion 2025-01-10 (Actual); Study Completion 2025-01-10 (Actual)

PRIMARY OUTCOMES:
SC and IV Arm: Area under the serum concentration-time curve from the pre-dose concentration extrapolated to infinity (AUCinf) | At predefined intervals throughout the study period (From Day 1 to Day 57)
  The concentration of anifrolumab in serum will be determined (AUCinf will be derived).
SC and IV Arm: Maximum observed serum (peak) concentration (Cmax) | At predefined intervals throughout the study period (From Day 1 to Day 57)
  The concentration of anifrolumab in serum will be determined (Cmax will be derived).
SC and IV Arm: Time to reach peak or maximum observed concentration (tmax) | At predefined intervals throughout the study period (From Day 1 to Day 57)
  The concentration of anifrolumab in serum will be determined (tmax will be derived).
SC and IV Arm: Area under the serum concentration-time curve from pre-dose concentration to time of last quantifiable concentration (AUClast) | At predefined intervals throughout the study period (From Day 1 to Day 57)
  The concentration of anifrolumab in serum will be determined (AUClast will be derived).
SC and IV Arm: half-life associated with the terminal slope of a semi-logarithmic concentration-time curve (t½λz) | At predefined intervals throughout the study period (From Day 1 to Day 57)
  The concentration of anifrolumab in serum will be determined (t½λz will be derived).
Bioavailability (F) | At predefined intervals throughout the study period (From Day 1 to Day 57)
  The concentration of anifrolumab in serum will be determined (F will be derived).
SC Arm: Apparent total body clearance of drug after extravascular administration (CL/F) | At predefined intervals throughout the study period (From Day 1 to Day 57)
  The concentration of anifrolumab in serum will be determined (CL/F will be derived).
SC Arm:Volume of distribution during the terminal phase after extravascular administration (Vz/F) | At predefined intervals throughout the study period (From Day 1 to Day 57)
  The concentration of anifrolumab in serum will be determined (Vz/F will be derived).
IV Arm: volume of distribution during the terminal phase after intravenous administration (Vz) | At predefined intervals throughout the study period (From Day 1 to Day 57)
  The concentration of anifrolumab in serum will be determined (Vz will be derived).
IV Arm: Apparent total body clearance of drug after intravenous administration (CL) | At predefined intervals throughout the study period (From Day 1 to Day 57)
  The concentration of anifrolumab in serum will be determined (CL will be derived).

SECONDARY OUTCOMES:
Adverse Event | From the time of signature of the ICF, throughout the study and including the follow-up period (approximately 12 weeks)
  Assessments related to AEs cover
  * Occurrence/frequency
  * Relationship to study intervention as assessed by investigator
  * Intensity
  * Seriousness
  * Death
  * AEs leading to discontinuation of study intervention
  * AESI
Vital Signs of blood pressure | From the time of signature of the ICF, throughout the study and including the follow-up period (approximately 12 weeks)
  * Observed value
  * Absolute change from baseline values over time
  * Vital sign status including change in abnormality (eg, low, normal, high) from baseline to minimum/maximum postbaseline value
  * Treatment-emergent changes outside predefined criteria
12-lead ECG measurements include heart rate, RR interval, PR interval, QRS duration, and QT interval | From the time of signature of the ICF, throughout the study and including the follow-up period (approximately 12 weeks)
  Assessments related to ECG cover:
  * Observed value
  * Absolute change from baseline values over time
  * ECG reading at baseline and each scheduled visit (normal, abnormal - clinically not significant, abnormal - clinically significant) including shifts in ECG interpretation compared to baseline
  * Treatment-emergent changes outside predefined criteria
Safety haematology laboratory parameters: WBC, Neutrophils absolute count, RBC, Lymphocytes absolute count, Hb, Monocytes absolute count, HCT, Eosinophils absolute count, MCV, Basophils absolute count, MCH, Platelets, MCHC, Reticulocytes absolute count | From the time of signature of the ICF, throughout the study and including the follow-up period (approximately 12 weeks)
  Assessments related to clinical laboratory safety
  * Observed value
  * Absolute change from baseline values over time
  * Laboratory status including change in abnormality (eg, low, normal, high) from baseline to minimum and maximum postbaseline value
  * Treatment-emergent changes in laboratory parameters outside predefined criteria Urinalysis categorisation as collected in the database including change in categorisation from baseline to the last post-baseline value.
Physical examination of height | From the time of signature of the ICF, throughout the study and including the follow-up period (approximately 12 weeks)
  Any new or aggravated clinically relevant abnormal medical finding at a physical examination as compared with the baseline assessment will be reported as an AE unless unequivocally related to the disease under study.
Vital Signs of pulse rate | From the time of signature of the ICF, throughout the study and including the follow-up period (approximately 12 weeks)
  * Observed value
  * Absolute change from baseline values over time
  * Vital sign status including change in abnormality (eg, low, normal, high) from baseline to minimum/maximum postbaseline value
  * Treatment-emergent changes outside predefined criteria
Vital Signs of body temperature | From the time of signature of the ICF, throughout the study and including the follow-up period (approximately 12 weeks)
  * Observed value
  * Absolute change from baseline values over time
  * Vital sign status including change in abnormality (eg, low, normal, high) from baseline to minimum/maximum postbaseline value
  * Treatment-emergent changes outside predefined criteria
Vital Signs of respiratory rate | From the time of signature of the ICF, throughout the study and including the follow-up period (approximately 12 weeks)
  * Observed value
  * Absolute change from baseline values over time
  * Vital sign status including change in abnormality (eg, low, normal, high) from baseline to minimum/maximum postbaseline value
  * Treatment-emergent changes outside predefined criteria
Safety clinical chemistry laboratory parameters: Sodium, CRP, Potassium, ALP, Urea, ALT, Creatinine, AST, Albumin, GGT, Calcium, TBL, Phosphate, Conjugated bilirubin, Glucose, Creatine kinase | From the time of signature of the ICF, throughout the study and including the follow-up period (approximately 12 weeks)
  Assessments related to clinical laboratory safety
  * Observed value
  * Absolute change from baseline values over time
  * Laboratory status including change in abnormality (eg, low, normal, high) from baseline to minimum and maximum postbaseline value
  * Treatment-emergent changes in laboratory parameters outside predefined criteria Urinalysis categorisation as collected in the database including change in categorisation from baseline to the last post-baseline value.
Safety urinalysis laboratory parameters: Glucose Protein, Blood, Microscopy (if positive for protein or blood) | From the time of signature of the ICF, throughout the study and including the follow-up period (approximately 12 weeks)
  Assessments related to clinical laboratory safety
  * Observed value
  * Absolute change from baseline values over time
  * Laboratory status including change in abnormality (eg, low, normal, high) from baseline to minimum and maximum postbaseline value
  * Treatment-emergent changes in laboratory parameters outside predefined criteria Urinalysis categorisation as collected in the database including change in categorisation from baseline to the last post-baseline value.
Physical examination of weight | From the time of signature of the ICF, throughout the study and including the follow-up period (approximately 12 weeks)
  Any new or aggravated clinically relevant abnormal medical finding at a physical examination as compared with the baseline assessment will be reported as an AE unless unequivocally related to the disease under study.
Physical examination of general appearance, the lungs, cardiovascular system, and the abdomen | From the time of signature of the ICF, throughout the study and including the follow-up period (approximately 12 weeks)
  Any new or aggravated clinically relevant abnormal medical finding at a physical examination as compared with the baseline assessment will be reported as an AE unless unequivocally related to the disease under study.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Wuhan, China

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org.
  Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/